CLINICAL TRIAL: NCT04682041
Title: Randomized Open-Label Clinical Study Evaluating the Impact of EnteraGam, a Nutritional Intervention Containing Bovine Plasma-Derived Immunoglobulin CoNcentrate, on Clinical Outcomes In People With COVID-19
Brief Title: Evaluating the Impact of EnteraGam In People With COVID-19
Acronym: PICNIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entera Health, Inc (Industry)
Collaborators: Lemus Buhils, SL (Unknown); Clinical Research Unit, IMIM (Hospital del Mar Medical Research Institute) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICNIC Study
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Coronavirus; Bovine Plasma-Derived Immunoglobulin
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized open-label clinical study evaluating the effectiveness of EnteraGam 10.0 g BID added to standard of care, as compared to standard of care alone, in subjects with COVID-19. Eligible subjects will be randomized in a 2:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EnteraGam + standard of care (Experimental): Subjects will receive EnteraGam® (oral nutritional therapy) + standard of care for COVID-19 for 2 weeks. Total study duration (including the screening phase) will be approximately 4 weeks.
  Interventions: Dietary Supplement: Bovine Plasma-Derived Immunoglobulin Concentrate; Other: Standard of care
- Control (standard of care) (Other): Subjects will receive standard of care for COVID-19 alone for 2 weeks. Total study duration (including the screening phase) will be approximately 4 weeks.
  Interventions: Other: Standard of care

INTERVENTIONS:
Dietary Supplement: Bovine Plasma-Derived Immunoglobulin Concentrate — EnteraGam® 10.0 g, containing 5.0 g of serum-derived bovine immunoglobulin/protein isolate (SBI) BID (every 12 hours) for 2 weeks.
  Other Names: EnteraGam®
  Arms: EnteraGam + standard of care
Other: Standard of care — Standard of care PSMAR protocol for COVID-19 patients.

SUMMARY:
Background:

Coronavirus Disease 2019 (COVID-19), caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), emerged as a potentially life-threatening disease in Wuhan, China, at the end of 2019. Since then, it has spread to almost 200 countries and infection rates are rapidly accelerating.

Overactivation of T cells resulting in immune dysfunction, dysfunction of the renin angiotensin system, and antibody-dependent enhancement are thought to contribute to the cytokine storm that results in acute respiratory distress syndrome (ARDS), culminating in death. In addition to causing respiratory symptoms, SARS-CoV-2 can cause diarrhea and has been isolated from the stool. SARS-CoV-2 binds to Angiotensin-converting enzyme 2 (ACE2) on lung alveolar type 2 cells, but ACE2 is also expressed in the absorptive enterocytes from the ileum and colon. The diarrhea may be caused by increased intestinal permeability due to binding of these receptors by the SARS-CoV-2.

Thus, an intervention to attenuate this cytokine storm may improve clinical outcomes in people with COVID-19. One such intervention is oral administration of serum bovine immunoglobulins, which decreases interleukin-6 (IL-6) levels safely with minimal side effects. Animal and human clinical studies have shown dietary supplementation with oral immunoglobulins improves mucosal immunity, specifically respiratory/pulmonary and GI mucosa, and decreases systemic inflammation, reducing the symptoms and severity of pulmonary inflammation and viral infections.

Hypothesis:

Dietary supplementation with EnteraGam® will decrease IL-6 levels and prevent disease progression in SARS-CoV-2 infected individuals.

Objectives:

To evaluate the effectiveness of the oral nutritional therapy EnteraGam® (serum-derived bovine immunoglobulin/protein isolate) to prevent disease progression of COVID-19 and to decrease IL-6 levels as compared to standard of care in subjects with COVID-19.

Methods:

Randomized open-label clinical study evaluating the effectiveness of EnteraGam® 10.0 g BID (every 12 hours) added to standard of care, as compared to standard of care alone, in subjects with COVID-19.

DETAILED DESCRIPTION:
Subject population:

Outpatient and inpatient male and non-pregnant females ≥18 years old, diagnosed with COVID-19 in the emergency department or admitted to the hospital but not requiring invasive mechanical ventilation or in the ICU.

Approximately 420 subjects will be randomized (2:1 ratio), 280 in the EnteraGam® arm and 140 in the control (standard of care) arm.

Nutritional intervention:

ImmunoLin is the active ingredient in EnteraGam®, a medical food developed and marketed by Entera Health in the US since 2013. ImmunoLin is an edible bovine plasma-derived immunoglobulin concentrate developed in 2001 as an immunoglobulin enriched plasma preparation for the human dietary supplement market. ImmunoLin is Generally Regarded as Safe (GRAS) following a letter of no objection from the US FDA in 2008. Physicians have prescribed EnteraGam® for patients with a variety of GI-related conditions.

Statistical methodology:

Efficacy: Based on per protocol analysis. Subjects lacking an assessment at Week 2 will be included in the analysis using the last available post-baseline data. Three pre-specified secondary analyses will be performed: 1) restricted to subjects with a comorbidity considered a major risk factor for hospitalization and disease severity (diabetes, cardiovascular disease, chronic lung disease, chronic renal disease, immunocompromised state); 2) restricted to age ≥ 50 years; 3) by inpatient only and outpatient only subgroups.

Additional analysis of covariance models with adjustment for Baseline characteristics and interactions may be examined in supportive or exploratory analyses.

Safety: All safety analyses will be based on all subjects who are randomized to EnteraGam and subsequently receive at least 1 packet of investigational product. Safety assessments will be analyzed by frequency of events/abnormalities for categorical values or summarized using descriptive statistics (mean, standard deviation, median, range, and number of observations).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Male or female. Females of childbearing (reproductive) potential must have a negative urine pregnancy test at screening.
3. Subject with diagnosis of COVID-19 based on + RNA or immunoglobulin M (IgM) test or compatible clinical presentation* who:

   1. is being discharged from the emergency department without hospitalization, or
   2. is admitted to the hospital or was previously hospitalized and still in the hospital, does not require invasive mechanical ventilation and does not require management in the intensive care unit. Inpatients can be enrolled in the study at any time of their hospitalization, if they comply with the inclusion criteria.

   (*)Compatible clinical presentation will consider compatible symptoms (cough, fever, myalgia, dyspnea, ageusia / anosmia) and examination of general condition, heart rate and respiratory rate, oxygen saturation, cardiopulmonary auscultation, compatible radiology.
4. Ability to consume EnteraGam.
5. Subject or surrogate decision maker is capable of understanding the requirements of the study, understands the language of the informed consent form, and is capable and willing to sign the informed consent form.

Exclusion Criteria:

1. Female subjects who are pregnant or breast-feeding.
2. Subject is enrolled in another randomized clinical trial.
3. Subject is taking anti-IL-6 treatment (e.g. tocilizumab), anti-IL-1 treatment (e.g. canakinumab, anakinra), or other biologic immunomodulators or immunosuppressant drugs. Note: Topical/inhaled immunomodulators and corticosteroids are not restricted.
4. Subject has immediate need for GI surgery or intervention for active GI bleeding, pancreatitis, peritonitis, intestinal obstruction, or intra-abdominal abscess.
5. Subject has active inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease, or celiac disease), GI malignancy, GI obstruction, pancreatitis, gastroparesis, carcinoid syndrome, amyloidosis, ileus, or cholelithiasis.
6. Subject has active gastric ulcer, duodenal ulcer, diverticulitis, colitis, enteritis, infectious gastroenteritis, or GI neoplasm, other than benign polyps.
7. Subject has a history of allergy or intolerance to beef or to any ingredient in the product.
8. Subject has active drug or alcohol abuse that in the opinion of the investigator may interfere with the subject's ability to comply with this protocol.
9. History of uncontrolled psychiatric disorders (includes significant depression or suicidal ideation), that in the opinion of the investigator may interfere with the subject's ability to comply with this protocol.
10. In the opinion of the investigator, progression to death is imminent and highly likely within the next 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma IL-6 levels | From baseline to Week 2
  Variation of IL-6 levels measured in plasma
COVID-19 disease progression by Week 2 | From baseline to Week 2
  Percentage of patients with COVID-19 who have disease progression by Week 2, defined as:
  1. For outpatients, return to emergency department for COVID-19 related manifestations or worsening of ≥1 level on the World Health Organization (WHO) 9-point ordinal scale.
  2. For inpatients, worsening of ≥1 level on the WHO 9-point ordinal scale.

SECONDARY OUTCOMES:
Change in dyspnea | At Week 2
  Variation of dyspnea presentation at Week 2 compared to baseline, assessed by daily symptoms questionnaire
Change in diarrhea | At Week 2
  Variation of diarrhea presentation at Week 2 compared to baseline, assessed by daily symptoms questionnaire
Change in fever | At Week 2
  Variation of fever presentation at Week 2 compared to baseline
Change in neutrophil count | At Week 2
  Variation of neutrophil count at Week 2 compared to baseline
Change in lymphocyte count | At Week 2
  Variation of lymphocyte count at Week 2 compared to baseline
Change in neutrophil/lymphocyte ratio | At Week 2
  Variation of neutrophil/lymphocyte ratio at Week 2 compared to baseline
Change in platelet count | At Week 2
  Variation of platelet count at Week 2 compared to baseline
Change in C-reactive protein | At Week 2
  Variation of C-reactive protein levels at Week 2 compared to baseline
Change in ferritin | At Week 2
  Variation of ferritin levels at Week 2 compared to baseline
Change in D-dimer | At Week 2
  Variation of D-dimer levels at Week 2 compared to baseline
Change in AST | At Week 2
  Variation of Aspartate Transaminase (AST/GOT) levels at Week 2 compared to baseline
Change in ALT | At Week 2
  Variation of Alanine Transaminase (ALT/GPT) levels at Week 2 compared to baseline
Time to worsening clinical status | From baseline to Week 2
  Time elapsed between baseline and disease progression, defined as:
  1. For outpatients, return to emergency department for COVID-19 related manifestations or worsening of ≥1 level on the WHO 9-point ordinal scale.
  2. For inpatients, worsening of ≥1 level on the WHO 9-point ordinal scale.

OTHER OUTCOMES:
Incidence of Adverse Events | From baseline to Week 2
  Incidence of serious and non-serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Güerri Fernández, MD, PhD, Principal Investigator — Hospital del Mar (Barcelona, Spain); Netanya S. Utay, MD, Principal Investigator — University of Texas Health Science Center at Houston (Houston, TX, USA)
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No